CLINICAL TRIAL: NCT06060093
Title: Effect of Ketone Ester Supplementation on Sleep and Recovery in Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Chiel Poffé, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S67089
Record Dates: First submitted 2023-08-29; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Ketosis; Hypoxia; Sleep
Keywords: Exercise; Ketones; Living-high Training-low
MeSH Terms: conditions — Ketosis; Hypoxia; Motor Activity | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: 1 session with both training and sleep in normoxia, supplemented with placebo (NPL)
  1 session with training in normoxia, sleep in hypoxia, supplemented with placebo (HPL)
  1 session with training in normoxia, sleep in hypoxia, supplemented with ketones (HKE)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normoxia - placebo (Placebo Comparator): Both training and sleep in normoxia, supplemented with placebo
  Interventions: Dietary Supplement: Placebo
- Hypoxia - placebo (Experimental): Training in normoxia and sleep in hypoxia, supplemented with placebo
  Interventions: Dietary Supplement: Placebo
- Hypoxia - ketones (Experimental): Training in normoxia and sleep in hypoxia, supplemented with ketones
  Interventions: Dietary Supplement: Ketone ester

INTERVENTIONS:
Dietary Supplement: Placebo — Water, 5% collagen(w/w), octoacetate (1 mM)
  Arms: Hypoxia - placebo; Normoxia - placebo
Dietary Supplement: Ketone ester — A total of 75g ketone ester supplementation will be administered in 3 bouts of 25g in order to establish intermittent exogenous ketosis: twice immediately after training, and one 30 minutes before sleep. The ketone ester used is (R)-3-hydroxybutyl (R)-3-hydroxybutyrate
  Arms: Hypoxia - ketones

SUMMARY:
This study specifically aims to elucidate the effects of IEK on sleep and recuperation in hypoxia, after training in normoxia. These conditions are in line with the widely applied live-high train-low strategy. Moreover, blood and tissue oxygenation status, as well as cerebral blood flow and cognitive function will be assessed.

DETAILED DESCRIPTION:
During training stages in order to prepare for an important event, sleep and recuperation are almost equally important as the appropriate training strategy. This training strategy often consists of living-high (sleeping at -stimulated- altitude) and training low (training at sea level). A decreased oxygen availability, also known as hypoxia, however often disrupts sleep quality and thus compromises the overall training efficiency. Ketones are recently found to improve sleep quality, thus potentially playing a pivotal role in altitude training. Therefore, the investigators want to evaluate the effects of ketones on sleep in hypoxia, after training in normoxia. Moreover, the effect on a performance test, during a simulated 30 min time trial on the next morning, will be investigated. During this protocol, cerebral blood flow will be assessed, as well as ventilation, blood and tissue oxygen status, heart rate variability, and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any experimental procedures
2. Males between 18 and 35 years old
3. Recreational or competitive cyclists performing regular cycling training sessions with an average training volume of more than 6 hours per week
4. Good health status confirmed by a medical screening
5. Body Mass Index (BMI) between 18 and 25
6. Normal sleep pattern as assessed by the Pittsburgh Sleep Quality Index
7. Moderate sleep chronotype (extreme morning and evening chronotypes will be excluded), assessed by the Horne and Östberg questionnaire

Exclusion Criteria:

1. Any kind of injury/pathology that is a contra-indication for hypoxic exposure and/or to perform high-intensity exercise, evaluated by a sport medical screening
2. Intake of any medication or nutritional supplement that is known to affect exercise, performance or sleep. Intake will be assessed during recruitment and the sport medical screening.
3. Intake of analgesics, anti-inflammatory agents, or supplementary anti-oxidants, from 2 weeks prior to the start of the study.
4. Recent residence or training under hypoxia; more than 7 days exposure to altitude > 1500m during the last 3 months preceding the study.
5. Night-shifts or travel across time zones in the month preceding the study
6. Blood donation within 3 months prior to the start of the study
7. Smoking
8. More than 3 alcoholic beverages per day
9. Pre-existing, diagnosed psychiatric conditions or diagnosed anxiety
10. Excessive daytime sleepiness as assessed by the Epworth scale
11. Depression or anxiety as assessed by the Beck Depression Inventory and Beck Anxiety Inventory. Only a score in the range of 'normal ups and downs' (score 1-10) for depression or 'minimal anxiety' (score 0-7) for anxiety are tolerated.
12. History of addiction or excessive caffeine/alcohol consumption assessed by a questionnaire
13. Any other argument to believe that the subject is unlikely to successfully complete the full study protocol

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Duration of different sleep stages | Throughout the entire duration of the night, up to 9 hours after individual bedtime
  Measured using polysomnography
Exercise performance | 30 minutes on the second morning of the protocol
  Measured as the average power output (W) during a 30 minutes time trial
Change in nocturnal oxygen saturation | Throughout the entire duration of the night, up to 9 hours after individual bedtime
  Measured using pulse oximetry
Absolute amount of nocturnal urinary catecholamine excretion | Subjects empty bladder before sleep and urine will be collected throughout the entire duration of the night, up to 9 hours after individual bedtime and in the morning immediately after waking up
  Measured using ELISA of collected nocturnal urine

CONTACTS AND LOCATIONS:
Overall Officials: Chiel Poffé, Dr., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stalmans M, Tominec D, Robberechts R, Lauriks W, Ramaekers M, Debevec T, Poffe C. A Single Night in Hypoxia Either with or without Ketone Ester Ingestion Reduces Sleep Quality without Impacting Next-Day Exercise Performance. Med Sci Sports Exerc. 2025 Apr 1;57(4):807-819. doi: 10.1249/MSS.0000000000003604. Epub 2024 Nov 18. PMID 39809236